CLINICAL TRIAL: NCT06586164
Title: Enhancing Rehabilitation for Veterans With Serious Mental Illness Via Biomarker-Informed Cognitive Training
Brief Title: Enhancing Rehabilitation for Veterans With Serious Mental Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5058-R; H230094 (Other: VA IRB)
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia; Psychosis; Serious Mental Illness; PTSD; Schizoaffective Disorder; Bipolar Disorder
Keywords: schizophrenia; psychosis; cognition; EEG; Serious mental illness; PTSD; Schizoaffective disorder; Bipolar disorder; clinical symptoms; function
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Stress Disorders, Post-Traumatic; Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to Targeted Cognitive Training (TCT) + Treatment as Usual (TAU) or Treatment as Usual (TAU)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TCT + TAU (Active Comparator): Subjects will complete 30 hours of Targeted Cognitive Training (TCT) in addition to their Treatment as Usual (TAU)
  Interventions: Behavioral: Targeted Cognitive Training
- TAU (No Intervention): Subjects will participate in their standard Treatment as Usual (TAU) PRRC program

INTERVENTIONS:
Behavioral: Targeted Cognitive Training — TCT is a computer-based cognitive training program in which participants train on progressively more difficult auditory processing exercises in order to improve speed, accuracy and fidelity of auditory information processing in order to generate gains in cognition and functioning.
  Other Names: TCT
  Arms: TCT + TAU

SUMMARY:
This study addresses the critical need for innovative therapeutic interventions in Veterans with serious mental illnesses (SMI) receiving care in VA Psychosocial Rehabilitation and Recovery Centers (PRRCs). The vast majority of individuals with SMI suffer from cognitive impairments, leading to chronic functional disability, and impaired outcomes, causing a significant strain on support networks and the VA healthcare system. This study aims to introduce an innovative mental health therapy, Targeted Cognitive Training (TCT), to Veterans struggling with serious mental illnesses (SMI). TCT works to improve basic sensory information processing and, ultimately, clinical, cognitive, and psychosocial functioning. By using EEG biomarkers to identify Veterans with SMI receiving care within VA Psychosocial Rehabilitation and Recovery Centers who are most likely to benefit from this treatment, and by understanding how best to implement this therapy, the investigators hope to enhance care and improve life quality for Veterans with SMI.

DETAILED DESCRIPTION:
This application addresses the critical need for innovative therapeutic interventions in Veterans with serious mental illnesses (SMI) receiving care in VA Psychosocial Rehabilitation and Recovery Centers (PRRCs). The vast majority of individuals with SMI suffer from cognitive impairments, leading to chronic functional disability, and impaired outcomes, causing a significant strain on support networks and the VA healthcare system. This application aims to introduce an innovative mental health therapy, Targeted Cognitive Training (TCT), to Veterans struggling with serious mental illnesses (SMI). TCT works to improve basic sensory information processing and, ultimately, clinical, cognitive, and psychosocial functioning.

TCT is a computerized intervention designed to sharpen the acuity and fidelity of sensory information processing through specific exercises that systematically increase demands on early perceptual and attentive processes. For many participants, TCT leads to "bottom-up" gains in perceptual functioning that lead to improvements in verbal learning and memory after 20-30h. While these benefits of TCT are evident at the group level, nearly half of all patients fail to show cognitive gains, even after extended 40-100h courses of TCT. By using EEG biomarkers to identify Veterans with SMI receiving care within VA Psychosocial Rehabilitation and Recovery Centers who are most likely to benefit from this treatment, and by understanding how best to implement this therapy, the investigators hope to enhance care and improve life quality for Veterans with SMI.

Enrolled patients complete clinical, cognitive and functional measures and candidate EEG biomarkers at baseline, and then are assigned to Treatment As Usual (TAU) vs. TCT+TAU arms (n=40/group) using stratified random sampling. TAU consists of participation in the standard PRRC programming that includes visits with PRRC clinicians, recovery coaching, groups and psychotherapy, peer services, and supported employment. Subjects randomized to TCT + TAU will also complete 30 hours of TCT consisting of three one-hour training sessions per week. Repeat assessment will occur after TCT session #10, 20 and 30 (or after the equivalent number of weeks have passed for TAU) and again 12 weeks after the cessation of TCT to evaluate the durability of observed gains.

This project will evaluate whether PRRC outpatients receiving 30 hours of TCT will exhibit significant improvements in clinical symptoms and cognition along with psychosocial functioning and quality of life compared with the TAU group. The investigators also hypothesize that favorable responses to 30 hours of TCT will be predicted by behavioral, cognitive, and EEG-based biomarkers measured at the beginning of the study. Finally the investigators will examine the acceptability of TCT and biomarker testing, as well as barriers and facilitators to implementation from the perspective of Veterans and PRRC clinicians based on feedback from study participants.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with SMI (e.g., schizophrenia, schizoaffective disorder, bipolar disorder, PTSD) being treated at PRRCs or co-located rehabilitative services.
* Age 18 and 83 years.
* Fluency in spoken and written English.
* Ability to detect 1000 Hz tones binaurally at a 40-dB sound pressure level.
* Ability to see with an acuity of 20/40 with both eyes tested together (corrected if applicable) by a standard printed Snellen eye chart reading card.

Exclusion Criteria:

* Estimated premorbid IQ below 70, as estimated via the WRAT-4 Reading subtest.
* Active substance use other than cannabis within the last 30 days as determined by CPRS review, self- report, or positive urine drug screen (obtained as part of the screening process).
* History of significant medical or neurological illness.
* Inability to comprehend or provide informed consent.

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Symptoms - Positive and Negative Syndrome Scale (PANSS) | 22 weeks
  Change from baseline clinical symptoms Positive and Negative Syndrome Scale (PANSS)
  The Positive and Negative Syndrome Scale (PANSS) will used to evaluate the presence, absence and severity of Positive, Negative and General Psychopathology symptoms of SZ. The PANSS is a 30-item scale arranged as 7 positive symptom subscale items, 7 negative symptom subscale items, and 16 general psychopathology symptom items. Each item has a definition and a basis for rating. All 30 items are rated on a 7-point scale (1=absent; 7=extreme). On the PANSS lower values are considered to be a better outcome.
Cognition - Matrics Consensus Cognitive Battery (MCCB) | 22 weeks
  Change from baseline cognition Matrics Consensus Cognitive Battery (MCCB) performance
  Change in Matrics Consensus Cognitive Battery (MCCB) performance from baseline is the outcome measure for cognition (using age- and gender-corrected T scores). The MCCB measures 7 cognitive domains: speed of processing, attention/vigilance, working memory (verbal and nonverbal), verbal learning, visual learning, reasoning/ problem solving and social cognition. MCCB verbal learning T-score is the primary cognitive outcome measure. Other MCCB domain T- scores will be used in secondary analyses. On the MCCB higher scores are indicative of better outcome.
Function - Functional Capacity: UCSD Performance-Based Skills Assessment, Brief Version (UPSA-B) | 22 weeks
  Functional Capacity will be assessed with the UCSD Performance-Based Skills Assessment, Brief Version (UPSA-B) at study entry and assessment intervals. The UPSA takes ~15 min to complete and incorporates role play to assess functional capacity in four broad domains: planning recreational activities, finances, communication and transportation. Raw scores on each subtest are transformed into a standardized subscale scores (0-25), which are summated to an overall
Function - Psychosocial Recovery: World Health Organization Disability Schedule 2.0 (WHODAS) | 22 weeks
  World Health Organization Disability Schedule 2.0 (WHODAS) will be used to assess psychosocial recovery. This detailed assessment consists of a 36-item questionnaire, where patients rate various aspects on a 5-point Likert scale. It covers six critical domains: cognition, mobility, self-care, social interactions, life activities, and societal participation. The WHODAS 2.0 will be used as an outcome measure for psychosocial recovery. Lower scores indicate better outcome on the WHODAS 2.0.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Light, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No